CLINICAL TRIAL: NCT05073718
Title: Efficacy of Low Dose Acetylsalicylic Acid in Preventing Adverse Maternal and Perinatal Outcomes in SARS-CoV-2 Infected Pregnant Women
Brief Title: SARS-CoV-2 and Acetylsalicylic Acid (SARA)
Acronym: SARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Hospital Universitario de Torrejón (Unknown); Hospital Universitario Infanta Leonor (Other); Hospital Sant Joan de Deu (Other); Hospital del Mar (Other); Eduardo Mondlane University (Other); Hospital Central de Maputo (Unknown); Hospital Geral de Mavalane (Unknown); Hospital Geral José Macamo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-000535-23
Record Dates: First submitted 2021-09-15; First posted 2021-10-11 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: SARS-CoV2 Infection; Covid19
Keywords: SARS-COV2; Acetylsalicylic acid; Asprin; ASA; COVID-19; Perinatal; Pregnancy
MeSH Terms: conditions — COVID-19 | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled multicentre clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study tablets will be identically packaged in small boxes. All study personnel, investigators and the participants will remain blinded throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDASA (n=200) (Experimental)
  Interventions: Drug: Low-dose acetylsalicylic acid
- Placebo (n=200) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose acetylsalicylic acid — In case of being positive for SARS-CoV-2 PCR or antigen test, she will be randomised 1:1 to receive daily LDASA (125 mg) or placebo, up to 36 weeks of pregnancy.
  Other Names: 125mg acetylsalicylic acid
  Arms: LDASA (n=200)
Drug: Placebo — Placebo
  Arms: Placebo (n=200)

SUMMARY:
SARS-CoV-2 infection in pregnancy is associated with an increased risk of adverse maternal and perinatal outcomes. One explanation is that the infection might increase the existing pregnancy-associated prothrombotic status, leading to a higher risk of placental and vascular complications. Administration of low-dose acetylsalicylic acid (LDASA) has shown to improve maternal and perinatal outcomes in women at high-risk of endothelial and placental complications. However, there are no data on the effect of LDASA in preventing complications in SARS-CoV-2- infected pregnant women. To reduce SARS-CoV-2- related complications in a highly vulnerable group to the infection, we will carry out this randomized, double-blind, placebo-controlled multicentre trial in 400 SARS-CoV-2-infected pregnant women. The study main objective is to evaluate the efficacy and safety of LDASA administered up to 36 weeks of gestation in SARS-CoV-2-infected pregnant women in reducing the incidence of adverse maternal and perinatal outcomes. Pregnant women tested positive up to 32 weeks of gestation with a SARS-CoV-2 rapid antigen or PCR test and agreeing to participate, will be randomised 1:1 to receive daily LDASA (125 mg) or placebo up to 36 weeks of gestation and be followed-up until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women up to 32 weeks of gestational age
* Aged 18 years or older*
* Willing to deliver at the recruitment health facilities

  * In Mozambique, in case of age below 18 years, the participant will be asked for the assent and the informed consent will be given by the legal tutor in accordance with the national regulations.

Exclusion Criteria:

* On regular ASA treatment for pre-eclampsia prevention
* On long-term non-steroidal anti-inflammatory medication
* Bleeding disorders, mainly haemophilia, hypoprothrombinaemia orVon Willebrand's disease
* History of hypersensitivity to ASA or to any of the excipients of the investigational product.
* History of peptic ulceration, including active, chronic or recurrent gastroduodenal ulcer; recurrent gastric discomfort History of gastric bleeding or perforation after treatment with aspirin or other non-steroidal anti-inflammatory drugs
* Inability to cooperate with the requirements of the study
* Severe COVID-19 disease (with any of the following: respiratory rate > 30 breaths/min; severe respiratory distress; SpO2 ≤ 93% on room air; acute respiratory distress syndrome; sepsis with acute organ dysfunction).
* Treatment resistant hyperemesis gravidarum
* Hypersensitivity to nonsteroidal anti-inflammatory drugs or to tartrazine (cross-reaction) or to any of the excipients used in its composition.
* Asthma.
* Severe renal or hepatic insufficiency.
* Nasal polyps associated with asthma that are induced or exacerbated by aspirin.
* Severe COVID-19 disease (with any of the following: respiratory rate > 30 breaths/min; severe respiratory distress; SpO2 ≤ 93% on room air; acute respiratory distress syndrome; sepsis with acute organ dysfunction).
* Treatment resistant hyperemesis gravidarum

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Rate of composite adverse maternal and perinatal adverse outcomes including miscarriage, foetal death, preeclampsia, maternal thromboembolic complications, placental abruption, preterm birth and small for gestational age. | up to 37 weeks

SECONDARY OUTCOMES:
Prevalence of SARS-CoV-2 infection and COVID-19 disease during pregnancy | up to 37 weeks
  maternal
Incidence of COVID-19-related admissions | up to 37 weeks
  maternal
Incidence of all-cause admissions | up to 37 weeks
  maternal
Incidence of all-cause outpatient attendances | up to 37 weeks
  maternal
Mean duration of symptoms-signs of COVID-19 | up to 37 weeks
  maternal
Frequency and severity of adverse events | up to 37 weeks
  maternal
Incidence of preeclampsia | up to 37 weeks
  maternal
Incidence of maternal thromboembolic complications and placental abruption | up to 37 weeks
  maternal
Maternal mortality rate | up to 37 weeks
  maternal
Incidence of histological placental abnormalities in SARS-CoV-2 infected pregnant women. | up to 37 weeks
  maternal
Prevalence of preterm birth (<37 weeks of gestational age) | up to 37 weeks
  embryo-foetal/infant
Prevalence of small for gestational age | up to 37 weeks
  embryo-foetal/infant
Prevalence of embryo and foetal losses (miscarriages and stillbirths) | up to 37 weeks
  embryo-foetal/infant
Frequency of congenital malformations | up to 37 weeks
  embryo-foetal/infant
Proportion of adverse perinatal outcome | up to 37 weeks
  embryo-foetal/infant
Neonatal morbidity | up to 37 weeks
  embryo-foetal/infant
Neonatal mortality rate | up to 37 weeks
  embryo-foetal/infant

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menéndez, Dr., Principal Investigator — Barcelona Institute for Global Health
Locations (4):
- Universidade Eduardo Mondlane, Maputo, Mozambique
- Spain (3):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Sant Joan de Déu, Barcelona, Catalonia
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818